CLINICAL TRIAL: NCT05605041
Title: Mindfulness in Medical Training: Using Headspace to Improve Sleep, Anxiety, and Burnout Among Resident Physicians
Brief Title: Mindfulness in Medical Training
Acronym: MiMT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough resources to proceed with the study
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000063
Record Dates: First submitted 2022-06-01; First posted 2022-11-04 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2022-07

CONDITIONS: Mindfulness, Burnout, Anxiety, Sleep
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Did Not Use Headspace (No Intervention): Those that did not use headspace during the time the study is conducted
- Did Use Headspace (Experimental): Those that were randomized into the group and used Headspace at least once during the study period
  Interventions: Device: Headspace

INTERVENTIONS:
Device: Headspace — Headspace is an app that allows users to practice mindfulness through guided meditation
  Arms: Did Use Headspace

SUMMARY:
Headspace, a smartphone application that provides guided meditation, mindfulness and sleep exercises, will be used as the intervention in improving sleep, anxiety, depression and burnout in all participating individuals selected from the University of Arizona College of Medicine-Tucson residents and fellows.

DETAILED DESCRIPTION:
The intervention of of daily meditation with the Headspace application will be used to determine if this is a possible effective intervention for decreasing the feeling of burnout. It is being proposed that it could improve the subjects' well-being both in the short-term and long term. The primary outcomes will be burnout, anxiety, depression and sleep. This study will use the Maslach Burnout Inventory to assess baseline burnout, as well as at 30 and 90 days post-intervention period. Sleep and anxiety and depression will be assessed using the Epworth Sleepiness Scale and Hospital Anxiety and Depression Scale (HADS) scores at the same intervals.

ELIGIBILITY:
Inclusion Criteria:

* University of Arizona resident or fellow

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
The Effects on Burnout | 30-90 days
  The intervention group will be asked to fill out the Maslachs Burnout Inventory (MBI) survey prior to intervention starting, 30 days after start of intervention and then again at 90 days after start of intervention). the MBI is a measure of three independent constructs - emotional exhaustion, depersonalization, and personal accomplishment. Lower scores will indicate less of an impact on those constructs. Higher scores indicate a stronger impact on those constructs. A score for emotional exhaustion includes anything <27, a low score is 0-18. For Depersonalisation a high score is anything >10 and a low score is 0-5. For Personal accomplishment a high score is 0-33 and low score is anything >40
The Effects on Sleep | 30-90 days
  The intervention group will be asked to fill out the Epworth Sleepiness Scale survey prior to intervention starting, 30 days after start of intervention and then again at 90 days after start of intervention). The scores will be analyzed to determine impact on sleep. Lower scores indicate a normal range of sleepiness, higher scores (18-24) will be indicative of severe sleepiness. Lower scores of 0-10 will be indicative of a normal range of sleepiness in healthy adults.
The effects on Anxiety and Depression | 30-90 days
  The intervention group will be asked to fill out the GAD-7 (Generalized Anxiety Disorder) questionnaire prior to intervention starting, 30 days after start of intervention and then again at 90 days after start of intervention. The scores will be analyzed to determine impact on anxiety and depression. Lower versus higher scores will be proportional to how much anxiety and depression that person is facing. A score of 0-4 is indicative of minimal anxiety and a score of > 15 is indicative of severe anxiety.

IPD SHARING:
Plan to Share IPD: Yes